CLINICAL TRIAL: NCT02091960
Title: A Phase 2, Multicenter, Open-label Study to Assess the Efficacy and Safety of Enzalutamide With Trastuzumab in Subjects With HER2+ AR+ Metastatic or Locally Advanced Breast Cancer
Brief Title: A Study to Assess the Efficacy and Safety of Enzalutamide With Trastuzumab in Patients With Human Epidermal Growth Factor Receptor 2 Positive (HER2+), Androgen Receptor Positive (AR+) Metastatic or Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9785-CL-1121; 2013-000093-29 (EudraCT Number)
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: HER2 Amplified; Advanced Breast Cancer; Human Epidermal Growth Factor Receptor 2 (HER2)
Keywords: Enzalutamide; Trastuzumab; Breast cancer; HER2; Androgen receptor positive; Xtandi
MeSH Terms: conditions — Breast Neoplasms | interventions — enzalutamide; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enzalutamide + Trastuzumab (Experimental): Participants received 160 mg enzalutamide orally once daily and 6 mg/kg trastuzumab administered by intravenous infusion or subcutaneous injection every 21 days. Participants continued on treatment until disease progression, unacceptable toxicity or any other discontinuation criteria were met.
  Interventions: Drug: Enzalutamide; Drug: Trastuzumab

INTERVENTIONS:
Drug: Enzalutamide — Capsules for oral administration
  Other Names: MDV3100; Xtandi
Drug: Trastuzumab — Intravenous infusion (IV) or subcutaneous injection if it is standard of care within a country
  Other Names: Herceptin

SUMMARY:
The purpose of this study was to evaluate the efficacy of enzalutamide with trastuzumab in patients with HER2+ AR+ metastatic or locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* The subject has histologically or cytologically proven adenocarcinoma of the breast that is HER2+
* The subject has AR+ breast cancer
* The subject has metastatic disease or has locally advanced disease that is not amendable to curative treatment
* The subject has measurable disease or nonmeasurable, evaluable disease per RECIST 1.1. (NOTE: pleural effusions, ascites or other third fluid space are not evaluable diseases per RECIST 1.1).
* The subject has received at least 1 line of therapy in the metastatic or locally advanced disease setting. The subject has been documented to have progressed by determination of the investigator on a regimen containing an anti-HER2 agent as the most recent regimen or the most recent anti-HER2 regimen was discontinued for any toxicity, with the exception of a cardiotoxicity.
* The subject has adequately recovered from toxicities due to prior therapy.
* The subject has an Eastern Cooperative Oncology Group performance (ECOG) status ≤ 1 at Screening and Day 1
* The subject has available at the site a representative, formalin-fixed, paraffin-embedded, tumor specimen that enabled the definitive diagnosis of breast cancer with adequate viable tumor cells in a tissue block (preferred) or ≥ 10 (20 preferred) freshly cut, unstained, serial slides and the associated pathology report

Exclusion Criteria:

* The subject has a severe concurrent disease, infection, or comorbidity that would make the subject inappropriate for enrollment.
* The subject has current or previously treated brain metastasis or active leptomeningeal disease. Brain imaging is required during screening in all subjects to exclude the presence of unequivocal central nervous system disease.
* The subject has a history of a non-breast cancer malignancy with the following exceptions:

  * The subject with a previous history of a non-invasive carcinoma is eligible if he/she has had successful curative treatment any time prior to Screening.
  * For all other malignancies, the subject is eligible if they have undergone potentially curative therapy and they have been considered disease free for at least 5 years prior to Screening.
* The subject has a history of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke, significant brain trauma).
* The subject has a history of loss of consciousness, cerebrovascular accident, or transient ischemic attack within 12 months before the Day 1 visit.
* The subject has had a hypoglycemic episode requiring medical intervention while on insulin (or other anti-diabetic) treatment within 12 months before Day 1.
* The subject had a major surgical procedure, substantial open biopsy, or significant traumatic experience within 28 days before the Day 1 visit, or anticipation of need for major surgical procedure during the course of the study.
* The subject has had palliative radiation therapy to bone metastases within 14 days prior to the Day 1 visit (side effects from radiation must be resolved).
* The subject has received chemotherapy, immunotherapy, or any other systemic anticancer therapy, with the exception of anti-HER2 therapy (e.g., trastuzumab), within 14 days prior to the Day 1 visit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (39):
- United States (16):
  - Site US10051, Anaheim, California
  - Site US10028, Los Angeles, California
  - Site US10035, San Francisco, California
  - Site US10079, Fort Myers, Florida
  - Site US10074, Gainesville, Florida
  - Site US10081, Chicago, Illinois
  - Site US10004, Indianapolis, Indiana
  - Site US10070, Boston, Massachusetts
  - Site US10078, St Louis, Missouri
  - Site US10072, Cincinnati, Ohio
  - Site US10048, Pittsburgh, Pennsylvania
  - Site US10029, Knoxville, Tennessee
  - Site US10042, Nashville, Tennessee
  - Site US10077, Nashville, Tennessee
  - Site US10076, Fort Worth, Texas
  - Site US10082, Houston, Texas
- Belgium (6):
  - Site BE32003, Edegem, Antwerp
  - Site BE32013, Brasschaat
  - Site BE32016, Brussels
  - Site BE32001, Charleroi
  - Site BE32009, Leuven
  - Site BE32007, Liège
- Canada (5):
  - Site CA15022, Ottawa, Ontario
  - Site CA15023, Toronto, Ontario
  - Site CA15028, Regina, Saskatchewan
  - Site CA15026, Saskatoon, Saskatchewan
  - Site CA15001, Québec
- Italy (6):
  - Site IT39005, Meldola, Forli
  - Site IT39008, Lecce
  - Site IT39003, Milan
  - Site IT39002, Milan
  - Site IT39001, Sondrio
  - Site IT39021, Udine
- Spain (3):
  - Site ES34014, Pozuelo de Alarcón, Madrid
  - Site ES34010, Barcelona
  - Site ES34013, Madrid
- United Kingdom (3):
  - Site GB44003, Edinburgh
  - Site GB44013, Manchester
  - Site GB44001, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Wardley A, Cortes J, Provencher L, Miller K, Chien AJ, Rugo HS, Steinberg J, Sugg J, Tudor IC, Huizing M, Young R, Abramson V, Bose R, Hart L, Chan S, Cameron D, Wright GS, Graas MP, Neven P, Rocca A, Russo S, Krop IE. The efficacy and safety of enzalutamide with trastuzumab in patients with HER2+ and androgen receptor-positive metastatic or locally advanced breast cancer. Breast Cancer Res Treat. 2021 May;187(1):155-165. doi: 10.1007/s10549-021-06109-7. Epub 2021 Feb 16. PMID 33591468
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14609&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 35 clinical sites in Belgium, Canada, Italy, Spain, the United Kingdom and the United States.
Pre-assignment Details: This study enrolled women with human epidermal growth factor receptor 2 positive (HER2+) and androgen receptor positive (AR+) metastatic or locally advanced breast cancer who progressed on anti-HER2 therapy in the metastatic or advanced setting.
Period: Overall Study
Arm/Group | Enzalutamide + Trastuzumab
Started | 103
Received Treatment | 103
Completed (Completed indicates participants with disease progression.) | 58
Not Completed | 45
Not completed — Death | 7
Not completed — Withdrawal by Subject | 1
Not completed — Miscellaneous Reasons | 37

BASELINE CHARACTERISTICS:
Arm/Group | Enzalutamide + Trastuzumab
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 98
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 90
  Race: Black or African American | 8
  Race: Asian | 3
  Race: American Indian or Alaskan Native | 0
  Race: Native Hawaiian or other Pacific Islander | 1
  Race: Other | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    Grade 0 | 51
    Grade 1 | 51
    Missing | 1
Time from Initial Diagnosis of Primary Cancer to Enrollment [Median (Full Range); unit: days] — Population: Participants for whom data were available
  days
    number analyzed (Participants) | 95
    (all) | 1199 [30 to 4713]
Histopathology at Diagnosis [Count of Participants; unit: Participants]
  Ductal | 73
  Inflammatory | 5
  Intraductal | 6
  Lobular | 6
  Mixed | 1
  Not otherwise specified | 1
  Other | 5
  Unknown | 6
Anatomic Stage [Count of Participants; unit: Participants] — Breast cancer staging is based on size of the tumor, whether cancer cells have spread to lymph nodes or to other parts of the body, how aggressive the cells appear when viewed under a microscope, whether the cancer cells have receptors for estrogen and progesterone or have a gene mutation that causes them to make excess HER2 protein, and the results of gene expression profiling tests. The stages of breast cancer range from 0 to IV, where Stage 0 is noninvasive or contained within the milk ducts and Stage IV breast cancer, also called metastatic, has spread to other areas of the body.
  Participants
    Stage 0 | 3
    Stage IA | 6
    Stage IB | 1
    Stage IIA | 14
    Stage IIB | 12
    Stage IIIA | 5
    Stage IIIB | 7
    Stage IIIC | 7
    Stage IV | 28
    Unknown | 20

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate was defined as the percentage of evaluable participants with best objective response of confirmed complete response or partial response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, or prolonged stable disease (≥ 24 weeks). Complete response (CR) was defined as the disappearance of all target and non-target lesions and no new lesions, and lymph nodes all < 10 mm in short axis. Partial response (PR) was defined as disappearance of target lesions or a ≥ 30% decrease in the size of target lesions, with persistence of non-target lesions and no new lesions. Stable disease (SD) was defined as < 30% decrease and < 20% increase in the size of target lesions, persistence of non-target lesions, and no new lesions. PR and CR required confirmation with equivalent or improved assessment no less than 4 weeks after the date that PR or CR was first observed. SD required confirmation with equivalent or improved assessment no less than 8 weeks after enrollment.
Time Frame: Tumor assessments were performed every 8 weeks through week 49, and then every 12 weeks thereafter until disease progression or death; the median duration of treatment was 70 days, and the maximum was 660 days.
Population: The efficacy evaluable set (EES) included all enrolled participants who had centrally assessed androgen receptor positive (AR+; defined as ≥ 10% of tumor cells with nuclear expression), received at least one dose of study drug, and had at least one available post baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Trastuzumab
Number analyzed (Participants) | 89
percentage of participants | 23.6 [15.2 to 33.8]

2. Secondary Outcome: Overall Response Rate at Week 24
Description: Overall response rate was defined as the percentage of evaluable participants with a best objective response of confirmed complete response (CR) or partial response (PR) per RECIST 1.1. Complete response was defined as the disappearance of all target and non-target lesions and no new lesions, and lymph nodes all < 10 mm in short axis. Partial response was defined as disappearance of target lesions or a ≥ 30% decrease in the size of target lesions with persistence of non-target lesions and no new lesions. PR and CR required confirmation with equivalent or improved assessment no less than 4 weeks after the date of scan that PR or CR was first observed.
Time Frame: 24 weeks
Population: Efficacy evaluable set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Trastuzumab
Number analyzed (Participants) | 89
percentage of participants | 3.4 [0.7 to 9.5]

3. Secondary Outcome: Best Overall Response Rate
Description: Best overall response was the best response across all time points, based on investigator assessments. Best overall response rate was defined as the percentage of evaluable participants with a best objective response of confirmed complete response (CR) or partial response (PR) at any time during the study per RECIST 1.1. Complete response was defined as the disappearance of all target and non-target lesions and no new lesions, and lymph nodes all < 10 mm in short axis. Partial response was defined as disappearance of target lesions or a ≥ 30% decrease in the size of target lesions with persistence of non-target lesions and no new lesions. PR and CR required confirmation with equivalent or improved assessment no less than 4 weeks after the date of scan that PR or CR was first observed.
Time Frame: as for outcome 1
Population: Efficacy evaluable set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Trastuzumab
Number analyzed (Participants) | 89
percentage of participants | 4.5 [1.2 to 11.1]

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the date of first dose of enzalutamide until the date of disease progression per RECIST 1.1, or death from any cause on study, whichever occurred first. Participants who initiated another antitumor therapy before documented progressive disease (PD) or death, or who progressed or died after missing 2 or more consecutive radiological assessments were censored at the date of the last radiological assessment showing no progression. Progressive disease was defined as a ≥ 20% increase in the size of target lesions and at least a 5 mm increase in size of target lesions from smallest size on study, or unequivocal progression of non-target lesions, or any new lesions.
Time Frame: From the date of first dose of study drug until disease progression or death; the median duration of treatment was 70 days, and the maximum was 660 days.
Population: Efficacy evaluable set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Enzalutamide + Trastuzumab
Number analyzed (Participants) | 89
days | 105.0 [61 to 116]

5. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time from the first date of enzalutamide treatment until the date of disease progression per RECIST 1.1. Participants who initiated another anti-tumor therapy before documented PD, who progressed after missing two or more consecutive radiological assessments or who died before disease progression were censored at the date of the last radiological assessment showing no progression.
Time Frame: as for outcome 4
Population: Efficacy analysis set
Measure: Median (Full Range); unit: days
Arm/Group | Enzalutamide + Trastuzumab
Number analyzed (Participants) | 89
days | 108.0 [61 to 116]

6. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the date of first documentation of response (CR or PR) until the date of disease progression per RECIST 1.1. Participants who initiated another anti-tumor therapy before documented PD, progressed after missing two or more consecutive radiological assessments or who died before disease progression were censored at the date of the last radiological assessment showing no progression.
Time Frame: as for outcome 1
Population: Efficacy evaluable set participants with a best overall response of CR or PR
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Enzalutamide + Trastuzumab
Number analyzed (Participants) | 4
days | NA [NA to NA] — Could not be estimated due to the low number of events

7. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from the first date of enzalutamide treatment to initial CR or PR and was calculated for participants with a CR or PR.
Time Frame: as for outcome 4
Population: Efficacy evaluable set with a best overall response of CR or PR
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Enzalutamide + Trastuzumab
Number analyzed (Participants) | 4
days | 57 [57 to 222]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered study drug/who underwent study procedures and did not necessarily have a causal relationship with treatment. Abnormalities identified during medical tests were defined as an AE if they induced clinical signs/symptoms, required active intervention, interruption or discontinuation of study medication, or were clinically significant to the investigator. An AE was defined as serious if any of the following resulted: Death, was life-threatening, persistent or significant disability/incapacity or substantial disruption of ability to conduct normal life functions, congenital anomaly/ birth defect, inpatient hospitalization/prolongation of hospitalization or other medically important event. TEAE was defined as an AE observed during the treatment emergent period, which is from first dose date of study drug to 30 days after last dose date or the start of subsequent treatment or date of death, whichever is first.
Time Frame: From the first dose date of study drug to 30 days after the last dose date of study drug or the start of subsequent treatment or date of death, whichever was first (Up to 3031 days)
Population: The Safety Analysis Set (SAF) which consisted of all participants who had received at least 1 or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide + Trastuzumab
Number analyzed (Participants) | 103
Participants
  Any treatment emergent adverse events (TEAE) | 97
  Enzalutamide Related TEAE | 75
  Trastuzumab Related TEAE | 40
  Any Drug Related TEAE | 78
  Deaths | 4
  Serious TEAE | 24
  Enzalutamide Related Serious TEAE | 3
  Trastuzumab Related Serious TEAE | 0
  Any Drug Related Serious TEAE | 3
  TEAE leading to discontinuation of enzalutamide | 23
  TEAE leading to discontinuation of trastuzumab | 21
  TEAE leading to discontinuation of any study drug | 24
  Discontinuation due to enzalutamide Related TEAE | 5
  Discontinuation due to trastuzumab Related TEAE | 5
  Discontinuation due to Any Drug Related TEAE | 9
  TEAE Leading to Dose Reduction | 7
  TEAE Leading to Dose Interruption | 23

ADVERSE EVENTS:
Time Frame: From the first dose date of study drug to 30 days after the last dose date of study drug or the start of subsequent treatment or date of death, whichever is first (Up to 3031 days).
Description: The Safety Analysis Set consisted of all participants who had received at least 1 or partial dose of study drug.
Arm/Group | Enzalutamide + Trastuzumab
All-Cause Mortality (participants affected / at risk) | 7/103
Serious Adverse Events (participants affected / at risk) | 24/103
Other Adverse Events (participants affected / at risk) | 89/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide + Trastuzumab (N=103)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (4)
Asthenia (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide + Trastuzumab (N=103)
Anaemia (Blood and lymphatic system disorders) | 9 (10)
Constipation (Gastrointestinal disorders) | 15 (16)
Diarrhoea (Gastrointestinal disorders) | 14 (16)
Dyspepsia (Gastrointestinal disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 28 (33)
Vomiting (Gastrointestinal disorders) | 10 (10)
Asthenia (General disorders) | 6 (6)
Fatigue (General disorders) | 37 (60)
Decreased appetite (Metabolism and nutrition disorders) | 15 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (16)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (14)
Dizziness (Nervous system disorders) | 14 (16)
Headache (Nervous system disorders) | 17 (19)
Restless legs syndrome (Nervous system disorders) | 7 (7)
Anxiety (Psychiatric disorders) | 9 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Hot flush (Vascular disorders) | 17 (18)
Hypertension (Vascular disorders) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT02091960/Prot_002.pdf
  • Statistical Analysis Plan (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT02091960/SAP_003.pdf